CLINICAL TRIAL: NCT05191563
Title: An Open-Label, Randomized, Single-Dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HCP1904 in Healthy Subjects
Brief Title: A Study to Compare the Pharmacokinetics, Safety and Tolerability Between Fixed-Dose Combination of HCP1904 and Co-Administration of RLD2001-2 and RLD2006 Tablets in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-CHOURS-101
Record Dates: First submitted 2021-07-05; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Reference-Test) (Experimental): Period 1: RLD2001-2 + RLD2006, Period2: HCP1904-1
  Interventions: Drug: HCP1904-1; Drug: RLD2006; Drug: RLD2001-2
- Sequence 2 (Test-Reference) (Experimental): Period 1:HCP1904-1, Period 2: RLD2001-2 + RLD2006
  Interventions: Drug: HCP1904-1; Drug: RLD2006; Drug: RLD2001-2

INTERVENTIONS:
Drug: HCP1904-1 — Take it once per period.
Drug: RLD2006 — Take it once per period.
Drug: RLD2001-2 — Take it once per period.

SUMMARY:
An Open-Label, Randomized, Single-Dose Crossover Study to Compare the Pharmacokinetics, Safety and Tolerability Between Fixed-Dose Combination of HCP1904 and Co-Administration of RLD2001-2 and RLD2006 Tablets in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who agree to use medically accepted dual contraceptives up to two months after the last administration date of the clinical trial drug and not to provide sperm.
4. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Cmax of Losartan | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
AUClast of Losartan | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
Cmax of EXP3174 | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
AUClast of EXP3174 | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
Cmax of Chlorthalidone | Day 1, Day 15: pre-dose(0 hour)~144hours
  Pharmacokinetic evaluation
AUClast of Chlorthalidone | Day 1, Day 15:pre-dose(0 hour)~144hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUC inf, Tmax, T1/2, Cl/F, Vd/F of Losartan | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
AUC inf, Tmax, T1/2, Cl/F, Vd/F of EXP3174 | Day 1, Day 15: pre-dose(0 hour)~48hours
  Pharmacokinetic evaluation
AUC inf, Tmax, T1/2, Cl/F, Vd/F of Chlorthalidone | Day 1, Day 15:pre-dose(0 hour)~144hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No